CLINICAL TRIAL: NCT01668771
Title: Self-Affirmation, Affect, and Implementation Intentions for Alcohol Cessation
Brief Title: Self-Affirmation and Response to Health Risk Information
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912162; 12-C-N162
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-05-13

CONDITIONS: Alcohol Drinking; Emotions; Ego
Keywords: Self-Affirmation; Affect; Alcohol
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Self-affirmation is the process of reflecting on values that a person considers important. This process may encourage people to be more open to information about health risks. It may also encourage them to change their behaviors or lifestyle to decrease these health risks. Researchers want to look at the effect of self-affirmation on people s responses to new health risk information. Because recent studies have linked alcohol consumption to increased risk of breast cancer, the study will focus on alcohol s link to breast cancer.

Objectives:

- To study how self-affirmation can change opinions following a message about a health risk.

Eligibility:

- Women at least 18 years of age who drink at least two alcoholic beverages per week and/or at least three alcoholic beverages per sitting.

Design:

* Participants will be recruited through an online panel. The study will be conducted entirely online.
* Participants will respond to two short studies. The first will ask about life events and how they make people feel. The second will look at how people respond to information about alcohol and breast cancer.
* For the first study, participants will write a paragraph or two about an important event in their lives. They will answer questions about how that event made them feel. They will also write a paragraph about an important personal value.
* For the second study, participants will read information about alcohol and breast cancer risk. They will then answer questions about this information. They will also answer questions about their beliefs about alcohol and breast cancer.
* Participants will receive financial compensation for being in this study.

DETAILED DESCRIPTION:
This study aims to examine whether emotional state moderates the effect of self-affirmation on intentions to engage in proactive behavior following a message about a health threat. Specifically, we propose to examine whether self-affirmation a process by which individuals reflect on cherished personal values differentially affects the persuasiveness of a message about the link between alcohol and breast cancer depending on whether individuals are in a particular emotional state. Previous evidence suggests that self affirmation may reduce defensiveness to threatening health information, increasing openness to the message and resulting in increased disease risk perceptions, disease-related worry, and intentions to engage in preventive behavior. However, self-affirmation may be differentially effective depending on the prior emotional state of the individual. Human subjects (women who report having consumed one or more alcoholic beverages in the past month) will be randomly assigned to write about an emotional event (something that made them happy, sad, angry, or hopeful) or to a neutral emotion condition (writing about a room in their house). Then, they will be randomly assigned to self-affirm (write about why a particular value is important to them) or to be in a control condition (write about why a particular value might be important to someone else). Following the autobiographical emotion task and self-affirmation, subjects will read about the link between alcohol and breast cancer. Finally, they will be asked a series of questions about their intentions to reduce drinking, their perceived risk of breast cancer, and their worry about breast cancer. Drawing on previous research, we hypothesize that self-affirmation will be most effective for those asked to recall a happy or angry experience, and least effective for those asked to recall a sad or hopeful experience

ELIGIBILITY:
* INCLUSION CRITERIA:
* Knowledge Networks panel respondents will be included if they are women who report having consumed the equivalent of 2-3 or more alcoholic beverage per week and/ or 3 or more alcoholic beverages in one sitting.
* Women will be included if they report drinking 3 or more drinks on any occasion, or more than 2-3 times per week.

EXCLUSION CRITERIA:

* Women will be excluded if they report never drinking alcohol or drinking monthly or 2-4 times per month, 1-2 drinks or less each time.
* All men, and women who report a lower threshold of alcohol consumption, will be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1116 (Actual)
Dates: Start 2012-08-11; Study Completion 2013-05-13

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Ferrer, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Armitage CJ, Harris PR, Hepton G, Napper L. Self-affirmation increases acceptance of health-risk information among UK adult smokers with low socioeconomic status. Psychol Addict Behav. 2008 Mar;22(1):88-95. doi: 10.1037/0893-164X.22.1.88. PMID 18298234
- [Background] Cavanaugh LA, Cutright KM, Luce MF, Bettman JR. Hope, pride, and processing during optimal and nonoptimal times of day. Emotion. 2011 Feb;11(1):38-46. doi: 10.1037/a0022016. PMID 21401223
- [Background] Crocker J, Niiya Y, Mischkowski D. Why does writing about important values reduce defensiveness? Self-affirmation and the role of positive other-directed feelings. Psychol Sci. 2008 Jul;19(7):740-7. doi: 10.1111/j.1467-9280.2008.02150.x. PMID 18727791